CLINICAL TRIAL: NCT03761641
Title: Pilot Study of NeuroTriage Device in Patients with Potential Brain Injury And/or Impairment
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jane Wigginton, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: 012015-030
Record Dates: First submitted 2015-10-19; First posted 2018-12-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Neurotriage — NeuroTriage binocular handset monitors pupil dynamics & eye position with infrared cameras. Rubber non-allergenic ocular spacers contoured to eye sockets come in contact with the face &cushion between the skin & eyepiece. During pupil dilation tests, an LED briefly illuminates the pupil. The NeuroTriage system measures neurological pupil index, constriction velocity, & dilation velocity. Total pupil dilation testing time is < 1 minute. During saccade-tracking tests, patients direct their gaze towards dim LED targets selectable across the range of view. Visual targets involve center-out ocular motion or smooth pursuit following of illusory movement. The NeuroTriage system measures eye position & movement velocity during these tests. Total saccade-tracking testing takes < 3 minutes. Ocular measures are non-invasive, are done quickly and commonly used to measure neurological function.

SUMMARY:
This protocol is aimed at collecting oculomotor response data from a variety of brain injuries and impairments, and to secondarily evaluate the functionality and ease of use of the NeuroTriage device in the ED in patients with any presumed brain injury and/or impairment. For example, prior studies in adolescents with a concussion have shown that they tend to overshoot the pattern when asked to follow the movement of the lights in the binoculars

DETAILED DESCRIPTION:
Study personnel will identify potential subjects in the ED, hospital and ICU during "peak hours" as appropriate through conferring with medical records, trauma logs, triage notes, and head CT, MRI, and other brain imaging orders as well as on-duty doctors and nurses to identify potential subjects. Many of the inclusion/exclusion criteria can be evaluated by a review of the potential subject's medical records, such as mechanism of injury or impairment, extent of non-head injuries, prior medical history, and prior clinical visits at the center of care. When a potential subject is identified and has been screened against the primary set of inclusion/exclusion criteria, they will be approached about the study.

Prior to enrolling a subject, the research personnel will screen the subject for competency to provide informed consent. This is necessary because, by its very nature, suspected brain injury patients may or may not be able to initially provide informed consent. The Galveston Orientation and Amnesia Test (GOAT) will be used as the standard assessment instrument for this screening. A score of 75 or greater on the GOAT would indicate that the subject is competent to provide informed consent. If the subject scores < 75 on the GOAT, then consent must be provided by a Legally Authorized Representative (LAR). This is a threshold of competency that has been used in previous studies here at UTSW.

Potential subjects that pass the GOAT will be given time to read the Consent Form and to consult with family members who may be present or by phone. If the subject agrees to participate, then they will sign the appropriate forms. A copy of the form will be given to the subject. The NeuroTriage and GOAT will then be serially performed on the patient no more than once every two hours (particularly in the ED, where the stay is often short) or with changes in neurological status.

ELIGIBILITY:
Criteria for Inclusion of Subjects:

One hundred individuals presenting to Parkland Emergency Department, Zale Lipshy and Clements Hospital for treatment diagnosed to be any form of mild, moderate or severe TBI, between the ages of 18 and 65 will be given the opportunity to participate in this study.

Patients injury should have occurred within the past 24 hours,and have an acute brain CT performed based on clinical care. We will enroll patients presenting to the Emergency Department (ED) with a history of TBI as per American Congress of Rehabilitation Medicine(ACRM) Criteria, in which the patient has sustained a traumatically induced* physiological disruption of brain function, as manifested by ≥ one of the following:

* Any period of loss of consciousness (LOC)
* Any loss of memory for events (e.g. amnesia) immediately before or after the accident-
* Any alteration of mental state at the time of the accident (feeling dazed, disoriented, and/or confused)
* Focal neurologic deficits that may or may not be permanent

Traumatically induced includes the head being struck, the head striking an object, or the brain undergoing an acceleration/deceleration movement (e.g. whiplash) without direct external trauma to the head.

All patients will need to be fluent in English or Spanish and be able to personally provide informed consent or have a legally authorized representative provide informed consent.

Individuals will not be excluded based on gender or race.

Criteria for Exclusion of Subjects:

Patients who have a penetrating Traumatic Brain Injury or a Spinal Cord Injury with ASIA score of C or worse will not be eligible for enrollment in this study.

* Any patients that are already participating in an interventional trial (e.g. drug, devise or behavioral) will be excluded.
* Non-English or Spanish speakers will be excluded.
* Any cognitive defect that limits comprehension of the study procedures and risks associated will be excluded.
* Patients with significant polytrauma that would interfere with assessments.
* Patients that have a significant history of pre-existing conditions that would interfere assessments (e.g.substance abuse, alcoholism, HIV/AIDS, major transmittable diseases that may interfere with consent, endstage cancers, learning disabilities, and developmental disorders).
* Patients on psychiatric hold or patients with a major debilitating mental health disorder (e.g. schizophrenia or bipolar disorder) will be excluded as they may interfere with follow-up and the validity of assessments.
* Patients with major debilitating neurological disease (e.g. stroke, CVA, dementia, tumor) impairing baseline awareness,cognition, or validity of follow-up and outcome assessment.
* Pregnancy in female subjects and prisoners in custody will be excluded.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to Parkland ED with suspected brain injury greater than 18 years of age, of an race or gender. Patients will need to be fluent in Spanish or English
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11-15 (Actual); Study Completion 2015-11-15 (Actual)

PRIMARY OUTCOMES:
Calibration of Neurotriage Device | Through study completion, 1 year
  Evaluate the number of rehabilitation device failure as reported by study team
Enjoyment of Neurotriage Device Use | Through Study Completion, 1 year
  Assess feasibility, ease of use and enjoyment for device in injured population. This will be measured by subject report. Subjects will verbally provide feedback as they use the software and hardware, changes will be made based on feedback received from participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jane G Wigginton, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No